CLINICAL TRIAL: NCT00041951
Title: Search for Genes Influencing Childhood Absence Epilepsy Study
Brief Title: Search for Genes Influencing Childhood Absence Epilepsy (CAE) Study
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 07-1441; R01NS037466 (NIH)
Record Dates: First submitted 2002-07-19; First posted 2002-07-22 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Absence Epilepsy; Epilepsy; Seizures
Keywords: Childhood Absence Epilepsy; CAE; Petit Mal; Epilepsy; Seizures; Genes; Inheritance; Genetics; Genetic Linkage
MeSH Terms: conditions — Epilepsy, Absence; Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CAE participants: Both parents and a child with CAE of families without other affected members (trios) or whole families with many members affected with epilepsy.
- Controls: Healthy individuals without epilepsy and no family history of epilepsy.

SUMMARY:
The purpose of our study is to identify gene(s) involved in the cause of childhood absence epilepsy (CAE).

DETAILED DESCRIPTION:
A high familial predisposition for epilepsy in patients with childhood absence epilepsy (CAE), also called petit mal epilepsy, suggests underlying genetic causes contributing to the disease. Several areas harboring potential absence epilepsy genes have been identified in the genome.

This study will further narrow down those areas and identify gene(s) involved in the cause of CAE by taking several approaches: 1. Comparing patients with CAE to healthy individuals without epilepsy and 2. Investigating whole families with many members affected with epilepsy).

Participation in this study requires an interview regarding medical and family history and saliva (spit) collection from all available family members of families with many epilepsy cases. For those families without a history of epilepsy, parents and children are asked to provide a small amount of saliva only. Healthy volunteers without epilepsy or a family history of seizures are asked to fill out an anonymous questionnaire and provide a small amount of saliva as well.

Although the study is based at Mount Sinai School of Medicine in New York, all study materials can be sent to your home at no cost to participants or their insurance. For the collection of saliva, special containers are provided and they can be shipped back to Mount Sinai in the pre-paid envelope provided. Study materials can be completed at your convenience.

Results from this study may enable scientists to understand the cause of absence seizures and, perhaps, other types of seizures as well and with this laying the foundation for better diagnosis and treatment of epilepsy patients in the future.

ELIGIBILITY:
Patients and their families:

Inclusion Criteria:

* Clinical diagnosis of classical (typical) Childhood Absence Epilepsy
* Good seizure control
* Must be able to give saliva sample

Exclusion Criteria:

* History of non-febrile seizures prior to the onset of typical absence seizures
* other neuropsychiatric or developmental disorders.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Whole families with many members affected with epilepsy or both parents and a child with CAE of families without other affected members (trios) and healthy individuals without epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 1998-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Saliva sample | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martina Durner, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States